CLINICAL TRIAL: NCT06600841
Title: Adebrelimab Combined with Non-platinum Chemotherapy and Fuzuloparib in the Treatment of Patients with Recurrent Platinum-resistant Ovarian Cancer (Sunrise Trial): a Single-Arm, Exploratory Study
Brief Title: Adebrelimab Combined with Non-platinum Chemotherapy and Fuzuloparib in Recurrent Platinum-resistant Ovarian Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Cancer Hospital (Other Government)
Collaborators: Fujian Provincial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SY-OC
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Platinum-resistant Ovarian Cancer (PROC); Immunotherapy
Keywords: Platinum-resistant Ovarian Cancer (PROC); adebrelimab; Fuzuloparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Immunotherapy group (Experimental): Drug: Adebrelimab, Non-platinum chemotherapy（Doxorubicin liposome/Paclitaxel-albumin/ or Gemcitabine）, fluzoparib Intervention：Adebrelimab plus Non-platinum chemotherapy（Doxorubicin liposome/Paclitaxel-albumin/ or Gemcitabine） induction therapy followed by maintenance therapy with adebrelimab plus fluzoparib.
  Interventions: Drug: Immunotherapy（Adebrelimab）

INTERVENTIONS:
Drug: Immunotherapy（Adebrelimab） — Adebrelimab plus non-platinum chemotherapy（Liposomal doxorubicin/Gemcitabine/ or nab-paclitaxel）and fluzoparib induction therapy followed by maintenance therapy with adebrelimab plus fluzoparib.
Drug: immunotherapy（Adebrelimab） — anti-PD-L1

SUMMARY:
The investigators explore the efficacy and safety of adebrelimab (PD-L1 inhibitor) plus Non-platinum chemotherapy and Fuzuloparib (PARP inhibitor) induction therapy followed by maintenance therapy with adebrelimab plus fluzoparib in platinum-resistant relapsed/metastatic ovarian cancer.

DETAILED DESCRIPTION:
Patients with platinum-resistant relapsed/metastatic ovarian cancer are treated with adebrelimab (PD-L1 inhibitor) plus Non-platinum chemotherapy and Fuzuloparib (PARP inhibitor) induction therapy for 6 cycles followed by maintenance therapy with adebrelimab plus fluzoparib

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70; Female;
2. Pathologically (including histologically) confirmed epithelial ovarian cancer, fallopian tube cancer, or primary peritoneal cancer (hereinafter referred to as ovarian cancer), recurrence within less than six months after the last treatment with platinum-containing chemotherapy;
3. Patients have at least one target lesion with measurable dimensions according to RECIST1.1 criteria;
4. HRR gene mutation confirmed by testing tissue or blood samples;
5. ECOG PS 0-1;
6. Major organ functions are normal and meet the following criteria:(1) Blood routine inspection standards must meet: (no blood transfusion within 14 days)a.HB≥100g/L, b. WBC≥3×10^9/L c. ANC≥1.5×10^9/L, d.PLT≥100×10^9/L; (2) Biochemical examination must meet the following standards: a. BIL ≤1.5 times the upper limit of normal (ULN); b. ALT and AST≤2.5×ULN, ALT and AST≤5×ULN in patients with liver metastases; c. Serum Cr≤1.5×ULN
7. Activated partial thromboplastin time (APTT) ≤ 1.5 times ULN, prothrombin time (PT) ≤ 1.5 times ULN, international normalized ratio (INR) ≤ 1.5 times ULN, unless the patient is receiving anticoagulation, as long as PT or APTT is within the expected range of anticoagulant use;
8. No severe heart, lung, liver or kidney disorders;
9. Women of childbearing age must have a pregnancy test (serum) within seven days before enrollment, have a negative result, and be willing to use appropriate methods of contraception during the trial period and eight weeks after the last administration of the test drug;
10. Estimated survival≥ 12 weeks;
11. Sign a written informed consent form and be able to comply with the visitation and related procedures set out in the program.

Exclusion Criteria:

1. Other clinical drug experiments in which other experimental research drugs are used concurrently with the study; 2. Patients with known hypersensitivity to fluzoparib or hypersensitivity to drug-active or inactive ingredients with a similar chemical structure to fluzoparib; 3. Patients with known hypersensitivity to adebrelimab or hypersensitivity to the active or inactive components of the drug having a similar chemical structure to adebrelimab; 4. Inability to swallow oral medications and any gastrointestinal disorders that may interfere with the absorption and metabolism of study medications, such as uncontrolled nausea and vomiting, gastrointestinal obstruction or malabsorption; 5. prior treatment with known or probable immune checkpoint inhibitors; 6. Have any active autoimmune disease or history of autoimmune disease (e.g., interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, myocarditis, nephritis, hyperthyroidism, hypothyroidism, including but not limited to these diseases or syndromes); Except vitiligo or recovered childhood asthma/allergies who do not require any intervention in adulthood; 7. Autoimmune-mediated hypothyroidism treated with stable doses of thyroid-replacement hormones; Type I diabetes mellitus with a stable dose of insulin; 8. A history of immunodeficiency, including a positive HIV test, or other acquired or congenital immunodeficiency disorders, or a history of organ transplantation and allogeneic bone marrow transplantation; 9. With unstable systemic diseases, such as hypertension that cannot be well controlled by antihypertensive drugs (systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥90 mmHg), severe arrhythmias, etc.; 10. Previous or current idiopathic pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonia, organising pneumonia, drug-induced pneumonia, or active pneumonia on screening-phase CT; 11. There are cardiac clinical symptoms or diseases that are not well controlled, such as: (1) cardiac insufficiency above NYHA grade 2 (2) unstable angina (3) acute myocardial infarction within 1 year (4) clinically significant supraventricular or ventricular arrhythmias requiring treatment or intervention (5) QTc>470ms; 12. Patients who are pregnant or breastfeeding, or who plan to become pregnant during study treatment; 13. The investigators considered it unsuitable for inclusion.

-

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate(ORR) | From the enrollment to the final documentation of response of the last subject (assessed up to 36 months)
  Objective Response Rate(ORR) was defined as the percentage of participants with the best (confirmed) overall response (BOR) of either CR or PR. ORR was assessed by the investigator according to RECIST version 1.1 and is based on BOR, defined as the best response recorded from the start of the study treatment until disease progression/recurrence or death. Participants needed two consecutive assessments of PR or CR to be responders. Only participants with measurable disease at baseline were included in the analysis of BOR, and those who did not have any evaluable post-baseline assessments were classified as not evaluable.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | From the enrollment to death, lost to follow-up, withdrawal, or study end, whichever occurred first, assessed up to 36 months
  PFS was defined as the time from randomization to first documented disease progression (PD) using Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1) or death from any cause, whichever occurred first. For target lesions, PD was defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum of the longest diameter recorded since treatment started or the appearance of 1 or more new lesions. For non-target lesions, PD was defined as the appearance of 1 or more new lesions and/or unequivocal progression of existing non-target lesions. The PFS will be will be estimated using Kaplan-Meier method. A Kaplan-Meier curve, median PFS, hazard ratio with appropriate confidence intervals will be reported.
Disease Control Rate(DCR) | From the enrollment to death, lost to follow-up, withdrawal, or study end, whichever occurred first, assessed up to 36 months
  DCR was defined as percentage of participants with best (confirmed) overall response (BOR) of either CR or PR or SD. DCR was assessed by the investigator according to RECIST version 1.1 and is based on BOR, which is defined as best response recorded from start of study treatment until disease progression/recurrence or death. Participants needed to have two consecutive assessments of PR or CR or SD to be a responder. Only participants with measurable disease at baseline were included in the analysis of BOR and who did not have any evaluable post-baseline assessments were classified as not evaluable.
Overall survival (OS) | From the enrollment to the death of last subject or the end of the clinical trial (assessed up to 36 months)
  defined as the time from the date of randomization to the date of death, regardless of the cause of death. Participants who were alive at the time of the analysis were censored at the date of the last follow-up assessment. Participants without follow-up assessment were censored at the day of last study medication and participants with no post-baseline information were censored at the date of randomization. The OS will be will be estimated using Kaplan-Meier method. A Kaplan-Meier curve, median OS, hazard ratio with appropriate confidence intervals will be reported.
Adverse events (AEs) | from the initiation of the first dose to 28 days after the last dose，assessed up to 36 months
  The incidence and severity of AEs, abnormalities in physical exams, vital sign assessments, clinical laboratory assessments

OTHER OUTCOMES:
Detection of PD-L1 expression level | 36 months
  Exploration outcome . Detection of PD-L1 expression level in tumor tissue by Immunohistochemistry
Detection of HRD status | 36 months
  Exploration outcome . Detection of HRD status in tumor tissue or peripheral blood by next-generation sequencing （NGS）.

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Cancer Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No